CLINICAL TRIAL: NCT02384109
Title: A Pharmacist-Coordinated Implementation of the Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kenrik Duru, Associate Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB#15-000310; R18DK105464-01 (NIH); IRB# 15-000310 (Other: UCLA OHRPP)
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Prediabetic State
MeSH Terms: conditions — Prediabetic State | interventions — Pharmacists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Pharmacist-coordinated shared decision making about treatment for pre-diabetes (lifestyle change and/or metformin), using a decision tool
  Interventions: Behavioral: Shared decision-making with pharmacists
- Usual Care (Placebo Comparator): Usual care for patients with a diagnosis of pre-diabetes
  Interventions: Other: Standard care from primary care providers

INTERVENTIONS:
Behavioral: Shared decision-making with pharmacists — Pharmacist will engage patient using Healthwise (TM) Decision Tool to help match their personal preferences and values with treatment options, specifically lifestyle change with a goal of 7% weight loss or metformin. Patients interested in lifestyle change will be referred to a CDC (Center for Disease Control and Prevention)-approved diabetes prevention program, and pharmacists will coordinate with primary care providers to prescribe metformin for patients interested in this treatment.
  Arms: Intervention
Other: Standard care from primary care providers — Primary care providers address pre-diabetes as part of usual care, which may involve no action, referrals, or treatment with medications.
  Arms: Usual Care

SUMMARY:
This proposed project will translate evidence-based strategies for diabetes prevention within the framework of an existing and highly utilized pharmacist-led diabetes care program. Our team includes investigators and practitioners with experience in implementing the DPP (Diabetes Prevention Program) as well as in community-based research. This proposal represents an opportunity to rapidly implement an innovative project addressing a critical area of significant unmet need, as the required key health system and community infrastructure are already in place. The intended outcome is the creation of a practical, effective and sustainable approach to increase evidence-based diabetes prevention strategies that can readily be adopted in other systems.

DETAILED DESCRIPTION:
The staggering number of Americans with prediabetes, now 1 in 3 adults,(1, 2) reinforces the urgency of implementing effective action to prevent incident diabetes. Several randomized controlled trials (RCTs) including the Diabetes Prevention Program (DPP) have demonstrated that both intensive lifestyle change and metformin significantly reduce the risk of progression to diabetes compared to placebo.(3-5) Prior efforts to disseminate treatment with lifestyle into practice have resulted in variable uptake and very limited population reach,(6) and their has been minimal to virtually no uptake of metformin for the treatment of prediabetes.

Within the University of California, Los Angeles (UCLA) Health System, the investigators have developed a program that embeds pharmacists in ambulatory clinics to co-manage patients with primary care physicians. The program, called Managing your Medications for Education and Daily Support (MyMEDS), has enrolled and treated almost 250 patients with diabetes and poorly-controlled cardiovascular risk factors in 14 primary care clinics over the last 12-months. Because of its effectiveness, leadership at UCLA Health has disseminated this program to all 28 primary care clinics in the system, and covers program-related costs including the pharmacists' salaries and appointment scheduling. The MyMEDS program is now part of routine clinical operations and represents a promising resource that could be mobilized to improve care for patients with prediabetes.

The investigators propose to implement a novel and pragmatic diabetes prevention intervention leveraging and extending the existing MyMEDS infrastructure. Within 10 of 20 randomly selected intervention clinics, the investigators will facilitate appointments for patients with prediabetes to the MyMEDS pharmacists. The pharmacists will educate patients about the DPP and engage them in shared decision-making about diabetes prevention, using a decision aid developed by HealthWise©. They will jointly develop a plan of care that includes intensive lifestyle change (preferred strategy since it has the greatest probability of reducing incident diabetes mellitus (DM)) and/or metformin, or take no immediate action and the pharmacist will communicate this decision to the primary care physician via our electronic health record (EHR). For participants who select lifestyle change, the investigators will partner with the YMCA (Young Men's Christian Association) of Metropolitan Los Angeles, which offers the DPP at multiple locations at sliding-scale rates. The YMCA will track attendance and participation in 16 weekly lifestyle change sessions and report this data to the pharmacists and study team (see Appendix 1 for letter of support). Patients can also participate in the UCLA DPP which is a separate DPP delivered on the UCLA campus. For patients who also select metformin, pharmacists will prescribe the medication as permitted under California law SB 493.(7) Pharmacists will see patients with prediabetes in routine follow-up to reinforce the care plan. This will be a pragmatic trial, and research funds will not be used to support delivery of the intervention. Rather than measuring the impact of lifestyle and/or metformin on incident diabetes or other clinical parameters, our primary endpoint will measure improvements in active engagement of treatment for prediabetes. The Specific Aims are as follows:

1. In a practice level, cluster-randomized, intention-to-treat trial, to test the effectiveness of using pharmacists to implement diabetes prevention strategies among patients with prediabetes, as compared to patients receiving usual care, on several outcomes with pre-planned stratification of a-e by age (<60 vs > 60 years):

   1. Uptake of intensive lifestyle change and/or metformin at 4 months (primary outcome)
   2. Proportion of patients who achieve >5% weight loss at 4 and 12 months
   3. Adjusted mean weight loss at 4 and 12 months, as a percentage of body weight at baseline
   4. Adjusted change in A1c at 12 months
   5. Adjusted change in systolic blood pressure at 12 months
2. To evaluate characteristics that will influence long-term sustainability of this intervention, among those in the intervention arm the investigators will measure:

   1. Acceptability to patients, physicians, pharmacists, clinic staff, and community partners including the YMCA
   2. Patient-reported psychosocial impact of their prediabetes, both positive and negative, stratified by the treatment selected
   3. Uptake of intensive lifestyle change and/or metformin at 4 months, by age (< 60 vs. 60+), gender, and race/ethnicity
   4. The incremental cost of program implementation per participant who successfully initiates lifestyle change and/or metformin.

I

ELIGIBILITY:
Inclusion Criteria:

* BMI (Body Mass Index) of >=24 (>=22 for Asians)
* Prediabetes based on A1c values of 5.7-6.4%

Exclusion Criteria:

* Any recorded A1c values of >6.5%
* ICD-9 billing codes of 250.xx
* Use of any antiglycemic medication
* Current or past participation in the Diabetes Prevention Program prior to providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 521 (Actual)
Dates: Start 2015-06; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Uptake of evidence-based diabetes prevention (lifestyle change or metformin) | 4 months
  Either attending 4/16 or 9/16 lifestyle change sessions, or taking metformin

SECONDARY OUTCOMES:
Weight change | 12 months
Change in A1c | 12 months
Change in systolic blood pressure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenrik Duru, MD, MSHS, Principal Investigator — University of California, Los Angeles
Locations (20):
- United States (20):
  - Toluca Lake Health Center, Burbank, California
  - 100 Medical Plaza Primary Care Suites 455 & 490, Los Angeles, California
  - Internal Medicine Women's Health Clinic Suites 250 & 290, Los Angeles, California
  - UCLA Internal Medicine Family Westwood Suite 465, Los Angeles, California
  - UCLA Internal Medicine Geriatrics Suite 365 & 420, Los Angeles, California
  - CPN Brentwood, Los Angeles, California
  - CPN West Washington Internal Medicine, Los Angeles, California
  - Pacific Palisades, Pacific Palisades, California
  - 12th Street Clinic, Santa Monica, California
  - Wilshire Office, Santa Monica, California
  - CPN Santa Monica 15th Street Family Medicine Practice, Santa Monica, California
  - CPN/Santa Monica Parkside, Santa Monica, California
  - Santa Moica Bay Physicians/20th Street 10th Floor, Santa Monica, California
  - Santa Monica Bay Physicians Plaza, Santa Monica, California
  - Santa Monica Bay Physicians/20th Street 3rd Floor, Santa Monica, California
  - Santa Monica Internal Medicine, Santa Monica, California
  - UCLA Family Health Clinic, Santa Monica, California
  - Santa Moica Bay Physicians Ocean Park, Santa Monica, California
  - Jack H. Skirball Health Center, Woodland Hills, California
  - CPN Woodland Hills Practice, Woodland Hills, California

REFERENCES:
- [Derived] Duru OK, Mangione CM, Turk N, Chon J, Fu J, Cheng G, Cheng F, Moss A, Frosch D, Jeffers KS, Castellon-Lopez Y, Tseng CH, Maranon R, Norris KC, Moin T. The Effectiveness of Shared Decision-making for Diabetes Prevention: 24- and 36-Month Results From the Prediabetes Informed Decision and Education (PRIDE) Trial. Diabetes Care. 2023 Dec 1;46(12):2218-2222. doi: 10.2337/dc23-0829. PMID 37770039
- [Derived] Moin T, Duru OK, Turk N, Chon JS, Frosch DL, Martin JM, Jeffers KS, Castellon-Lopez Y, Tseng CH, Norris K, Mangione CM. Effectiveness of Shared Decision-making for Diabetes Prevention: 12-Month Results from the Prediabetes Informed Decision and Education (PRIDE) Trial. J Gen Intern Med. 2019 Nov;34(11):2652-2659. doi: 10.1007/s11606-019-05238-6. Epub 2019 Aug 30. PMID 31471729